CLINICAL TRIAL: NCT03917407
Title: U01 Pilot Trial of DUR-928 in Patients With Moderate and Severe Alcoholic Hepatitis
Brief Title: DUR-928 in Patients With Alcoholic Hepatitis
Acronym: DUR-928/AH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Craig James McClain (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor-Investigator, Craig James McClain, Professor, University of Louisville
Organization: University of Louisville (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19.0776; 1U01AA026934-01 (NIH)
Record Dates: First submitted 2019-03-27; First posted 2019-04-17 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Alcoholic Hepatitis
Keywords: Alcoholic Hepatitis; Alcoholic Liver Disease
MeSH Terms: conditions — Hepatitis, Alcoholic; Liver Diseases, Alcoholic | interventions — 25-hydroxycholesterol 3-sulfate

STUDY DESIGN:
Intervention Model Description: An Open-Label, Dose Escalation Study to Assess the Safety, and Pharmacodynamics signals of DUR 928 in Patients with AH. DUR-928 will be administered in 100 mL 5% dextrose or 0.9% sodium chloride by slow intravenous infusion over 2 hrs (50mL/h) until entire dose is given at Day 1 and Day 4. If a patient meets the hospital discharge criteria prior to the 2nddose, the patient will receive only one dose of DUR-928 instead of 2 doses.
Masking Description: Dur-28 treated moderate AH: 7 Dur-28 treated severe AH: 12 Observational AH: 8 Steroid Treated AH: 16
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm1: DUR-928 treatment for moderate alcoholic hepatitis (Active Comparator): Enrolled alcoholic hepatitis patients would have MELD of 11-20; and have met inclusion and exclusion criteria. DUR-928 as a novel study treatment would be administered in patients with moderate alcoholic hepatitis (AH) as determined by the absence of suspected unexpected serious adverse reaction (SUSAR).
  Interventions: Drug: DUR-928 (Moderate AH)
- Arm 2: DUR-928 treatment for severe alcoholic hepatitis. (Active Comparator): Enrolled alcoholic hepatitis patients would have MELD of 21-30; and have met inclusion and exclusion criteria. DUR-928 as a novel study treatment would be administered in patients with severe alcoholic hepatitis (AH) as determined by the absence of suspected unexpected serious adverse reaction (SUSAR).
  Interventions: Drug: DUR-928 (Severe AH)

INTERVENTIONS:
Drug: DUR-928 (Moderate AH) — A total of no more than two doses of DUR-928 will be given, with 72 hrs between each dose. A second dose of the assigned study treatment (test drug) will be repeated 3 days after Dose 1 to patients who are still hospitalized. If a patient meets the discharge criteria prior to Day 4, the patient will receive only one dose of DUR 928.
  Patients of Part A (MELD 11-20) will follow the dose escalation procedure based on cohort; each patient will receive an intravenous infusion dose of:
  * Cohort 1A: 30 mg of DUR-928in 100 mL 5% dextrose or 0.9% sodium chloride administered over approximately 2 hrs via IV infusion.
  * Cohort 2A: 90 mg of DUR 928 in 100 mL5% dextrose or 0.9% sodium chloride administered over approximately 2 hrs via IV infusion.
  * Cohort 3A: 150 mg of DUR 928 in 100 mL5% dextrose or 0.9% sodium chloride administered over approximately 2 hrs via IV infusion.
  Other Names: Sulfated oxysterol: 5 cholesten-3β, 25-diol 3-sulfate (25HC3S)
  Arms: Arm1: DUR-928 treatment for moderate alcoholic hepatitis
Drug: DUR-928 (Severe AH) — Dose escalation to the next cohort will be determined after review of safety, tolerability and pharmacokinetic data of the previous cohort. Dose escalation for Part B will follow the same requirements as for Part A. The dose levels for Part B are planned to be the same as Part A.
  Patients of Part B (MELD 21-30) will follow the dose escalation procedure based on cohort; each patient will receive an intravenous infusion dose of:
  * Cohort 1B: 30 mg of DUR-928 in 100 mL 5% dextrose or 0.9% sodium chloride administered over approximately 2 hrs via IV infusion.
  * Cohort 2B: 90 mg of DUR 928 in 100 mL5% dextrose or 0.9% sodium chloride administered over approximately 2 hrs via IV infusion.
  * Cohort 3B: 150 mg of DUR 928 in 100 mL5% dextrose or 0.9% sodium chloride administered over approximately 2 hrs via IV infusion More details on preparation and administration of study drug will be provided in the Investigation Product Manual for this study.
  Other Names: Sulfated oxysterol: 5 cholesten-3β, 25-diol 3-sulfate (25HC3S)
  Arms: Arm 2: DUR-928 treatment for severe alcoholic hepatitis.

SUMMARY:
The proposed study is An Open-Label, Dose Escalation Study to Assess the Safety, and Pharmacodynamics (PD) signals of DUR 928 in Patients with AH. DUR-928 will be administered in 100 mL 5% dextrose or 0.9% sodium chloride by slow intravenous infusion over 2 hrs (50mL/h) until entire dose is given at Day 1 and Day 4. If a patient meets the hospital discharge criteria prior to the 2nd dose, the patient will receive only one dose of DUR-928 instead of 2 doses.

DETAILED DESCRIPTION:
The study will be conducted in 2 Parts using a staggered parallel design. Part A will include patients with MELD scores of 11-20, and Part B will include patients with MELD of scores 21-30.

Within each Part, the study will be conducted using a starting dose level of 30 mg with sequential dose escalation following review of safety results of the prior dose level by the sponsor, the principal investigators. The planned subsequent doses of DUR-928 after the starting dose are 90 mg and 150 mg.

Patients with a MELD score of 21-30 (Part B) receiving the 30 mg dose level will only be enrolled once safety review of the 30 mg dose of DUR-928 in patients with MELD score 11-20 (Part A) has been completed. The subsequent dose escalation in Part B will not proceed until the sponsor, and the principal investigators, and the medical monitor complete the review of safety of the 30 mg dose level and determine it is safe to do so.

At each dose level within a Part, 4 patients will be treated. If no SUSAR is observed, dose escalation to the next dose cohort within the Part will proceed. If 1 of the 4 patients demonstrates a SUSAR in a given dose level, an additional 2 patients will be treated at that dose level. If only 1 of the 6 patients demonstrates SUSAR, the next cohort of four patients will enter at the next dose level. If 6 patients are dosed and 2 or more demonstrate SUSAR at that dose level, the study will deescalate to a lower dose (but higher than the previous dose). At subsequent dose levels, the maximum tolerated dose (MTD) is defined as the dose level where no more than 1 of 6 patients experiences a SUSAR.

If no SUSAR is observed, dose escalation to the next dose cohort will proceed. All patients will be followed up to Day 28 (Total duration of patient engagement is 33 days).

Trial Population:

Patients with AH will be enrolled at Louisville associated hospitals in the US. The target number of participants to complete the study is 24-36. During the trial, patients should receive standard of care as determined by the PI (e.g. pentoxifylline or corticosteroids).

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent (either from patient or patient's legally acceptable representative)
2. Male or female patients 21 years of age or older with BMI ≥ 20 to ≤ 40 kg/m2
3. Patients with alcoholic hepatitis defined as:

   1. History of heavy alcohol abuse: > 40 g/day in females or > 60 g/day in males for a minimum period of 6 months, AND
   2. Consumed alcohol within 12 weeks of entry into the study, AND
   3. Serum bilirubin > 3 mg/dL AND AST > ALT, but less than 300 U/L AND
   4. MELD score between 11-30, inclusive
4. No evidence of active infection as determined by the investigator. If infection is initially suspected clinically,

   1. blood cultures, urine cultures, and peritoneal cultures should be without growth for 48 hrs, AND
   2. peritoneal cell count should be less than 250 Polymorphonuclear cell (PMN)/ml. If infection is diagnosed, then the infection must be

   <!-- -->

   1. treated with antibiotics, AND
   2. documented negative blood cultures for 48 hrs, or for spontaneous bacterial peritonitis (SBP) 25% reduction in PMN count prior to enrollment.
5. Women of child-bearing potential (defined as females who are not surgically sterile or who are not over the age of 52 and amenorrheic for at least 12 months) must utilize appropriate birth control throughout the study duration. Acceptable methods that may be used are abstinence, birth control pills ("The Pill") or patch, diaphragm, intrauterine device (IUD/ coil), vaginal ring, condom, surgical sterilization or progestin implant or injection, or sexual activity limited to a sterile (e.g., vasectomized) male partner.
6. Male patients must agree to use a medically acceptable method of contraception/birth control throughout the study duration.

Exclusion Criteria:

1. Other or concomitant cause(s) of liver disease as a result of:

   1. Autoimmune liver disease (positive anti-mitochondrial antibody and smooth muscle antibody, positive reading on anti-nuclear antibody titer > 1:160)
   2. Wilson disease (ceruloplasmin levels < 10 mcg/L)
   3. Vascular liver disease
   4. Drug induced liver disease
   5. Surface antigen positive hepatitis B (HBsAg+). Note: patients with isolated core antibody (HBcAb) are not excluded.
   6. Acute hepatitis A
   7. Acute HCV or chronic hepatitis C with a history of decompensated cirrhosis. Note: patients with stable chronic Hep C Virus (HCV) or successfully treated HCV are not excluded.
2. Co-infection with human immunodeficiency virus (HIV)
3. Positive Urine Drug Screen (amphetamines, barbiturates, benzodiazepines, cocaine and opiates) except THC and legal prescription medications.
4. Any active malignancies other than curatively treated skin cancer (basal cell or squamous cell carcinomas) or any other malignancy diagnosed within the last five years
5. Active tuberculosis on chest x-ray at study entry
6. Significant systemic or major illness other than liver disease, including coronary artery disease, cerebrovascular disease, pulmonary disease, renal failure, serious psychiatric disease, that, in the opinion of the Investigator would preclude the patient from participating in and completing the study
7. Patients requiring the use of vasopressors or inotropic support. Prior use of inotropic support will be allowed if the condition has stabilized within the first 7 days of admission to the hospital
8. Liver biopsy, if carried out, showing findings not compatible with AH
9. Any patient that has received any investigational drug or device within 30 days of dosing or who is scheduled to receive another investigational drug or device at any time during the study
10. Patients who are taking drug products that are primarily the substrates of CYP2C8, such as chloroquine, paclitaxel, rosiglitazone, repaglinide
11. If female, known pregnancy, or has a positive serum pregnancy test, or is lactating/breastfeeding
12. Serum creatinine > 2.5 mg/dL
13. Patients who have had organ transplantation (such as liver, kidney, lung, heart, bone marrow, or stem cell etc.), other than cornea transplant
14. Stage 3 or greater encephalopathy by West Haven criteria

Ages: 21 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-09-24 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Assessment of Treatment-Emergent Adverse Events | 4.5 years.
  Assess the safety and tolerability of DUR-928 in patients with alcoholic hepatitis (AH) as determined by the absence of suspected unexpected serious adverse reaction (SUSAR).
Pharmacodynamic signals of DUR-928: Model for End-Stage Liver Disease [MELD] | 33 days.
  Drivers of the Model for End-Stage Liver Disease [MELD] score individually using a formula (3.78×ln[serum bilirubin (mg/dL)] + 11.2×ln[INR] + 9.57×ln[serum creatinine (mg/dL)] + 6.43 that incorporates following lab measures: International Normalized Ratio [INR], and Serum Creatinine and Serum Total Bilirubin [units for both: mg/dl]) at baseline, Day 7 and Day 28. Participant's involvement in study: 33 days maximum.
Pharmacodynamic signals of DUR-928: Liver Biochemical Biomarker "Alanine Aminotransferase" | 33 days.
  Improvement in liver biochemistry at baseline, Day 7 and Day 28 (Alanine Aminotransferase [ALT, unit: IU/L]. Participant's involvement in study: 33 days maximum.
Pharmacodynamic signals of DUR-928: Liver Biochemical Biomarker "Aspartate Aminotransferase" | 33 days.
  Improvement in liver biochemistry at baseline, Day 7 and Day 28 for Aspartate Aminotransferase [AST, unit: IU/L]. Participant's involvement in study: 33 days maximum.
Pharmacodynamic signals of DUR-928: Liver Biochemical Biomarker "Total Bilirubin" | 33 days.
  Improvement in liver biochemistry at baseline, Day 7 and Day 28 for Total Bilirubin [unit: mg/dl]. Participant's involvement in study: 33 days maximum.
Pharmacodynamic signals of DUR-928: Liver Biochemical Biomarker "Albumin" | 33 days.
  Improvement in liver biochemistry at baseline, Day 7 and Day 28 for Albumin [unit: g/L]. Participant's involvement in study: 33 days maximum.
Quality of life biomarkers: 36-item Short Form Survey (SF-36). | 33 days.
  Quality of Life biomarkers (eg. SF-36) at Baseline, Day 7 and Day 28. Participant's involvement in study: 33 days maximum.
Biomarkers of liver cell death: Cytokeratin 18 (CK18) | 33 days.
  Novel liver cell death markers: Cytokeratin18M65 (K18M65), and Cytokeratin18M30 (K18M30). Units: IU/L. Evaluation at baseline, day 7 and day 28. Participant's involvement in study: 33 days maximum.
Biomarkers of Inflammation (Interleukins): Interleukin 6 and Interleukin 8 | 33 days.
  interleukin 6 (IL6, unit: pg/mL) and Interleukin 8 (IL8, unit: pg/mL) at baseline, day 7 and day 28. Participant's involvement in study: 33 days maximum.
Biomarkers of Inflammation: C-reactive Protein | 33 days.
  C-reactive Protein (CRP, unit: mg/dL) assessed at baseline, day 7 and days 28. Participant's involvement in study: 33 days maximum.

CONTACTS AND LOCATIONS:
Overall Officials: Vatsalya Vatsalya, M.D., Study Director — Department of Medicine, University of Louisville; Craig J McClain, M.D., Principal Investigator — Department of Medicine, University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make Individual patient data (IPD) available.

REFERENCES:
- [Result] Liangpunsakul S. Clinical characteristics and mortality of hospitalized alcoholic hepatitis patients in the United States. J Clin Gastroenterol. 2011 Sep;45(8):714-9. doi: 10.1097/MCG.0b013e3181fdef1d. PMID 21085006
- [Result] Menon KV, Gores GJ, Shah VH. Pathogenesis, diagnosis, and treatment of alcoholic liver disease. Mayo Clin Proc. 2001 Oct;76(10):1021-9. doi: 10.4065/76.10.1021. PMID 11605686
- [Result] FDA, Draft guidance for Drug Interaction Studies. February 2012.
- [Result] Orman ES, Odena G, Bataller R. Alcoholic liver disease: pathogenesis, management, and novel targets for therapy. J Gastroenterol Hepatol. 2013 Aug;28 Suppl 1(0 1):77-84. doi: 10.1111/jgh.12030. PMID 23855300
- [Result] O'Shea RS, McCullough AJ. Treatment of alcoholic hepatitis. Clin Liver Dis. 2005 Feb;9(1):103-34. doi: 10.1016/j.cld.2004.11.004. PMID 15763232
- [Result] Thursz MR, Richardson P, Allison M, Austin A, Bowers M, Day CP, Downs N, Gleeson D, MacGilchrist A, Grant A, Hood S, Masson S, McCune A, Mellor J, O'Grady J, Patch D, Ratcliffe I, Roderick P, Stanton L, Vergis N, Wright M, Ryder S, Forrest EH; STOPAH Trial. Prednisolone or pentoxifylline for alcoholic hepatitis. N Engl J Med. 2015 Apr 23;372(17):1619-28. doi: 10.1056/NEJMoa1412278. PMID 25901427